CLINICAL TRIAL: NCT01333384
Title: A Non-Interventional Retrospective (12 Months) and Prospective (at Least 24 Months) Resource Utilization Study, in the Population of Polish Acromegalic Patients Treated With Somatuline Autogel at Normal (4 Weeks) or Extended (6 or 8 Weeks) Dosing Interval
Brief Title: Study in Polish Acromegalic Patients Treated With Somatuline Autogel
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-38-52030-739
Record Dates: First submitted 2011-04-08; First posted 2011-04-12 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate over the 24 month prospective follow up - in everyday clinical practice - resource utilization and effectiveness of the treatment of acromegalic patients in Poland with Somatuline Autogel 120 mg including extended injection intervals.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with acromegaly treated for at least three injections with Somatuline Autogel 120 mg
* Subjects must be treated for acromegaly for at least 1 year, with medical treatment prior to inclusion. One year historical data must be available

Exclusion Criteria:

* Active participation in any interventional or any other non-interventional acromegaly clinical study. Previous participation in observational / post-marketing study of other somatostatin analogue should not be an exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Observation of 150 patients out of 500 routinely treated with somatostatin analogues in Poland
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Percentage variation of Insulin-like growth factor-1 (IGF-1) levels | 24 months

SECONDARY OUTCOMES:
Mean growth hormone (GH) levels | 24 months
Proportion of patients with GH levels below 1.0 microgram/liter | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Ipsen Central Contact, Warsaw, Poland